CLINICAL TRIAL: NCT00464490
Title: A Prospective, Randomized, Controlled Study on the Use of Dexmedetomidine to Facilitate Extubation in Surgical Intensive-Care-Unit Patients Who Failed Previous Weaning Attempts
Brief Title: Use of Dexmedetomidine to Facilitate Extubation in Surgical ICU Patients Who Failed Previous Weaning Attempts
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of eligible participants
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0703054
Record Dates: First submitted 2007-04-19; First posted 2007-04-23 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Intubation; Difficult; Respiration Disorders
Keywords: Weaning; Extuvation; Dexmedetomidine
MeSH Terms: conditions — Respiration Disorders | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Hospital Ventilation Weaning Protocol (No Intervention): Control. Hospital weaning protocol
- Dexmedetomidine for Extubation (Experimental): Dexmedomidine infusion to facilitate extubation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine .5mcg/kg/hr-.7mcg/kg/hr 1hour prior to extubation. Dexmedetomidine will be titrated according to blood pressure, RASS and heart rate response and the dose will be lowered only after sedation is discontinued or markedly reduced.
  Other Names: Precedex
  Arms: Dexmedetomidine for Extubation

SUMMARY:
Mechanical ventilation commonly is associated with patient agitation requiring sedation to alleviate discomfort and reduce excessive central respiratory drive. Upon recovery from acute respiratory failure, sedation is reduced to facilitate the withdrawal of ventilatory support. In some patients, abrupt reduction in sedation provokes severe agitation that causes catecholamine release resulting in severe hypertension, tachycardia and tachypnea. This requires increased sedation to bring hemodynamic and respiratory function under control.

Dexmedetomidine is an alpha-2 receptor agonist with both sedative and analgesic properties that allows for the reduction in the anesthetic and analgesic requirements in the perioperative setting. In addition to its sedative effects, alpha-2 receptor stimulation in the central nervous system inhibits sympathetic activity and reduces plasma epinephrine and norepinephrine levels, thereby lowering both arterial blood pressure and heart rate. Because alpha-2 receptor stimulation does not cause respiratory depression, dexmedetomidine may facilitate the transition to unassisted breathing in profoundly agitated patients. The investigators will prospectively evaluate dexmedetomidine in 30 patients who could not be extubated because of agitation with hemodynamic instability and tachypnea.

The purpose of this study is to test if a larger prospective randomized controlled pilot study can show that dexmedetomidine facilitates weaning and extubation in patients who have failed previous attempts because of agitation and hyperdynamic cardiopulmonary response.

DETAILED DESCRIPTION:
Sixty patients who are admitted to the surgical intensive care unit (ICU) at San Francisco General Hospital will be referred to the investigators for enrollment into a prospective, unblinded, randomized study of dexmedetomidine. Each patient will be considered by the critical care team as a suitable candidate for weaning and extubation based on inclusion/ exclusion criteria. Pregnant patients will not be enrolled and this will be determined by a negative urine or serum pregnancy test from admission. If none is available a pregnancy test will be performed prior to enrollment. Patients considered difficult to wean will be based on the following criteria:

Eligible patients will be randomized to either the control arm or the dexmedetomidine arm in a 1:1 ratio by using sealed envelopes.

Patient randomized to the control arm will be extubated per standard hospital protocol. This arm of the study will be observational and these patients will be extubated by the attending physician for that patient whenever they are hemodynamically stable enough to tolerate another weaning trial. The study team will collect the same data points for the control arm as in the dexmedetomidine arm. This includes ABGs, heart rate, mean blood pressure, respiratory rate and RASS scores (see description below of data points and collection time points.) Arterial blood gases will be drawn for the control arm of the study.

Patients on the dexmedetomidine arm will be started on dexmedetomidine at either 0.5 mcg/kg/hr or 0.7 mcg/kg/hr 1 hour prior to extubation. The drug calculation was based upon an average taken between the patient's measured and predicted body weight. Background sedation will be generally facilitated with lorazepam, midazolam or propofol, while analgesia will be maintained with either fentanyl or hydromorphine. After starting dexmedetomidine background sedation and analgesia will be titrated down and discontinued if possible. Analgesia levels also will be reduced if tolerated. Dexmedetomidine will be titrated according to blood pressure, RASS and heart rate response and the dose will be lowered only after sedation is discontinued or markedly reduced. Aerosolized lidocaine (20 mg) therapy will be initiated prior to the weaning trial to prevent excessive coughing in all patients.

Shortly after the dexmedetomidine infusion is started, PSV will be commenced at 5 cm H2O above 5 cm H2O of continuous positive airway pressure (CPAP). Patients will be weaned to CPAP and evaluated for extubation.

1.) Arterial blood gases will be obtained in all patients with an arterial line at three points in time: just prior to dexmedetomidine infusion, during the CPAP trial, and approximately 30 minutes after extubation.

3.) Heart rate, mean blood pressure, RASS, and respiratory rate will be collected at fifteen minute intervals 1 hour prior to dexmedetomidine infusion, during the 1 hour infusion of dexmedetomidine prior to the extubation then 5, 15, 30, 45, 60, 90 and 120 minutes after extubation for a total of 4 hours of data collection.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than 70 years old
2. Normothermia (36.5 degrees centigrade)
3. Normal sinus rhythm
4. Hemodynamically stable (systolic blood pressure [SBP] > 110 mmHg)
5. Ejection fraction (EF) > 40%/absence of congestive heart failure (CHF)
6. Cardiac index > 2.5 L/min/m2
7. Minimal inotropic support (< 3 mcg/kg/min dobutamine)
8. Adequate coagulation profile
9. Adequate urine output (> 100 ml/hr)
10. Primary service and critical care physician agreement

Exclusion Criteria:

1. Prior use of clonidine or alpha-antagonists
2. Prior history of intravenous drug abuse (IVDA) or alcohol abuse (ETOH)
3. Evidence of heart block
4. Difficulty with oxygenation/ventilation
5. Renal or hepatic insufficiency
6. Pregnant (positive urine or serum pregnancy test upon admission)
7. Patient received dexmedetomidine > 24 hours

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-11; Primary Completion 2012-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julin F Tang, M.D., M.S., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total accrual reached 42 of the planned 60; unanticipated common usage of Dexmedetomidine led to difficulty recruiting intubated/sedated patients who had not used it within protocol-specified period prior to enrollment. Also, some providers were not willing to allow patient assignment to the control arm given the popular usage of the drug.
Groups:
- Dexmedetomidine for Extubation (DG): Dexmedomidine infusion to facilitate extubation
  Dexmedetomidine: Dexmedetomidine .5mcg/kg/hr-.7mcg/kg/hr 1hour prior to extubation. Dexmedetomidine titrated according to blood pressure, RASS and heart rate response and the dose lowered only after sedation was discontinued or markedly reduced.
- Standard Hospital Protocol (CG): Control. Standard hospital weaning protocol
Period: Overall Study
Arm/Group | Dexmedetomidine for Extubation (DG) | Standard Hospital Protocol (CG)
Started | 21 | 21
Completed | 10 | 10
Not Completed | 11 | 11
Not completed — Physician Decision | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine for Extubation (DG) | Standard Hospital Protocol (CG) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Ramsay Sedation Scale (RSS) [Mean (Standard Deviation); unit: units on a scale] — The RSS defines the conscious state from a level 1: the patient is anxious, agitated or restless, through the continuum of sedation to a level 6: the patient is completely unresponsive.
  units on a scale | 3.5 (1.2) | 2.1 (1.1) | 3 (3)

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Ventilation Time
Time Frame: time from first weaning attempt to successful extubation
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dexmedetomidine for Extubation (DG) | Standard Hospital Protocol (CG)
Number analyzed (Participants) | 10 | 10
hours | 59.2 (139.4) | 203.9 (150.7)
Statistical Analysis 1: Comparison: Dexmedetomidine for Extubation (DG) vs Standard Hospital Protocol (CG); H(0): Ventilator time (DG) = Ventilator time (CG); Test type: Superiority or Other; p = 0.02, t-test, 2 sided — P-value <0.05 was considered significant

ADVERSE EVENTS:
Time Frame: 2 hour pre- to 2 hours post-extubation
Description: We monitored for adverse events associated with the study intervention.
Groups:
- Standard Hospital Protocol (CG): Control. Hospital weaning per standard protocol
Arm/Group | Dexmedetomidine for Extubation (DG) | Standard Hospital Protocol (CG)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Lower than anticipated enrollment due to unwillingness of providers to assign patients to the control group led to smaller-than-planned samples for analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes